CLINICAL TRIAL: NCT00715624
Title: A Randomized, Double-blind, Placebo-controlled, 2-arm Parallel-group, Multicenter Study With a 24-week Main Treatment Period and an Extension Assessing the Efficacy and Safety of AVE0010 in Patients With Type 2 Diabetes Insufficiently Controlled With Basal Insulin
Brief Title: GLP-1 Receptor Agonist Lixisenatide in Patients With Type 2 Diabetes for Glycemic Control and Safety Evaluation, on Top of Basal Insulin
Acronym: GETGOAL-L
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC6016; 2007-005886-36 (EudraCT Number)
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: hyperglycemia, GLP-1, metformin, insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Insulin Resistance | interventions — lixisenatide; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide (Experimental): 2-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
  Interventions: Drug: Lixisenatide (AVE0010); Drug: Basal Insulin; Drug: Metformin; Device: Pen auto-injector
- Placebo (Placebo Comparator): 2-step initiation regimen of volume matching placebo: 10 mcg QD for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
  Interventions: Drug: Placebo; Drug: Basal Insulin; Drug: Metformin; Device: Pen auto-injector

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Lixisenatide
Drug: Placebo — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Placebo
Drug: Basal Insulin — Dose to be kept stable.
Drug: Metformin — Metformin if given to be continued at stable dose (1.5 gram per day) up to the end of treatment.
Device: Pen auto-injector
  Other Names: OptiClik®

SUMMARY:
The purpose of this study is to evaluate the benefits and risks of lixisenatide (AVE0010), in comparison to placebo, as an add-on treatment to basal insulin with or without metformin over a period of 24 weeks of treatment, followed by an extension.

The primary objective is to assess the effects of lixisenatide when added to basal insulin on glycemic control in terms of glycosylated hemoglobin (HbA1c) reduction at Week 24.

The secondary objectives are to assess the effects of lixisenatide when added to basal insulin on body weight, 2-hour postprandial plasma glucose (PPG) after standardized meal challenge test, percentage of patients reaching HbA1c less than 7 percent (%), percentage of patients reaching HbA1c less than or equal to 6.5%, fasting plasma glucose (FPG), change in 7-point self-monitored plasma glucose (SMPG) profiles, change in basal insulin and total insulin doses; to evaluate safety, tolerability, pharmacokinetics (PK) and anti-lixisenatide antibody development.

DETAILED DESCRIPTION:
Patients who complete the 24-week main double-blind treatment would undergo a variable double-blind extension treatment, which ends for all patients at approximately the scheduled date of Week 76 visit (Visit 25) for the last randomized patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed for at least 1 year before screening visit, insufficiently controlled with basal insulin with or without metformin

Exclusion Criteria:

* HbA1c less than (<) 7 % or greater than (>) 10% at screening
* At the time of screening age < legal age of majority
* Pregnant or breastfeeding women or women of childbearing potential with no effective contraceptive method
* Type 1 diabetes mellitus
* Treatment with basal insulin for less than 3 months prior to screening or insulin regimen changed during the last 3 months prior to screening
* Basal insulin dose at screening <30 units/day and/or not at a stable dose (+/- 20 percent [%]) during the last 2 months
* If treatment with metformin, no stable dose of at least 1.5 gram/day (except for South Korea: at least 1.0 gram/day) for at least 3 months prior to screening visit
* FPG at screening >250 milligram per deciliter (mg/dL) (>13.9 millimole per liter [mmol/L])
* History of hypoglycemia unawareness
* Body mass index less than or equal to (<=) 20 kilogram per square meter (kg/m^2)
* Weight change of >5 kg during the 3 months preceding the screening visit
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, or inflammatory bowel disease
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within 3 months prior to the time of screening
* Within the last 6 months prior to screening, history of myocardial infarction, stroke, or heart failure requiring hospitalization
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Cardiovascular, hepatic, neurological, endocrine disease, active malignant tumor or other major systemic disease or patients with short life expectancy making implementation of the protocol or interpretation of the study results difficult, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting systolic blood pressure (SBP) or diastolic blood pressure (DBP) >180 millimeter of mercury (mmHg) or >95 mmHg, respectively
* Laboratory findings at the time of screening: aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase: >2 times upper limit of the normal (ULN) laboratory range; amylase and/or lipase: >3 times ULN; total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome); hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100 000/mm^3; positive test for Hepatitis B surface antigen and/or Hepatitis C antibody and positive serum pregnancy test in females of childbearing potential
* Any clinically significant abnormality identified on physical examination, laboratory tests, electrocardiogram, or vital signs at the time of screening that, in the judgment of the investigator or any sub-investigator, precludes safe completion of the study or constrains efficacy assessment
* Patients who are considered by the investigator or any sub-investigator as inappropriate for this study for any reason (for example, impossibility to meet specific protocol requirements, such as attending scheduled visits, being able to do self-injections; likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol; investigator or any sub-investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol)
* Use of other oral or injectable antidiabetic or hypoglycemic agents other than metformin or basal insulin (for example, sulfonylurea, alpha-glucosidase inhibitor, thiazolidinedione, rimonabant, exenatide, dipeptidyl-peptidase-4 inhibitors, fast-acting insulin for 1 week or more) within 3 months prior to the time of screening
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 1 week or more within 3 months prior to the time of screening
* Any previous treatment with lixisenatide or participation in any previous study with lixisenatide
* Use of any investigational drug within 3 months prior to study
* Renal impairment defined with creatinine >1.4 mg/dL in women and creatinine >1.5 mg/dL in men (applicable only for patients with metformin treatment)
* End-stage renal disease as defined by a calculated serum creatinine clearance of <15 milliliter/minute and/or patients on dialysis, if no treatment with metformin
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to gastroparesis and gastroesophageal reflux disease requiring medical treatment, within the previous 6 months
* History of allergic reaction to any glucagon like peptide-1 (GLP-1) agonist in the past (for example, exenatide, liraglutide) or to metacresol
* Additional exclusion criteria at the end of the run-in phase: informed consent withdrawal; lack of compliance during the single-blind placebo run-in phase (>2 injections missed); and patient with any adverse event which precludes the inclusion in the study, as assessed by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2008-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, San Juan, Puerto Rico
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] Riddle MC, Aronson R, Home P, Marre M, Niemoeller E, Miossec P, Ping L, Ye J, Rosenstock J. Adding once-daily lixisenatide for type 2 diabetes inadequately controlled by established basal insulin: a 24-week, randomized, placebo-controlled comparison (GetGoal-L). Diabetes Care. 2013 Sep;36(9):2489-96. doi: 10.2337/dc12-2454. Epub 2013 Apr 29. PMID 23628617
- [Derived] Yao J, Zhang M, Zhang X, Zhang J. Impact of Type 2 Diabetes Duration on the Efficacy and Safety of Add-on Lixisenatide in Asian Individuals Receiving Basal Insulin: A Pooled Analysis. Diabetes Ther. 2023 Apr;14(4):653-669. doi: 10.1007/s13300-023-01369-6. Epub 2023 Feb 21. PMID 36809495
- [Derived] Davidson JA, Stager W, Paranjape S, Berria R, Leiter LA. Achieving postprandial glucose control with lixisenatide improves glycemic control in patients with type 2 diabetes on basal insulin: a post-hoc analysis of pooled data. Clin Diabetes Endocrinol. 2020 Jan 14;6:2. doi: 10.1186/s40842-019-0088-5. eCollection 2020. PMID 31956422
- [Derived] Charbonnel B, Bertolini M, Tinahones FJ, Domingo MP, Davies M. Lixisenatide plus basal insulin in patients with type 2 diabetes mellitus: a meta-analysis. J Diabetes Complications. 2014 Nov-Dec;28(6):880-6. doi: 10.1016/j.jdiacomp.2014.07.007. Epub 2014 Jul 18. PMID 25130920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 111 centers in 15 countries between July 29, 2008 and February 8, 2011. The overall duration of treatment was at least 76 weeks (24 weeks main double-blind treatment; variable double-blind extension treatment).
Pre-assignment Details: A total of 879 patients were screened of which 383 (43.6%) were screen failures; main reason for screen failure was glycosylated hemoglobin (HbA1c) values being out of the defined protocol range (greater than or equal to 7% and less than or equal to 10%). A total of 496 patients were randomized.
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo: 10 microgram (mcg) once daily (QD) subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
- Lixisenatide: 2-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
Period: Overall Study
Arm/Group | Placebo | Lixisenatide
Started | 167 (Randomized) | 329
Treated/Safety Population | 167 (All patients who were exposed to at least 1 dose, regardless of amount of treatment administered.) | 328
Modified Intent-to-Treat(mITT)Population | 166 (All patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment.) | 327
Completed | 115 | 213
Not Completed | 52 | 116
Not completed — Adverse Event | 12 | 37
Not completed — Lack of Efficacy | 11 | 11
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 11 | 25
Not completed — Familial and personal reasons | 10 | 22
Not completed — Poor compliance | 6 | 13
Not completed — Sponsor decision | 0 | 4
Not completed — Incorrect randomization (not treated) | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to the end of treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lixisenatide | Total
Number analyzed (Participants) | 167 | 328 | 495
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (9.8) | 57.4 (9.5) | 57.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 182 | 267
  Male | 82 | 146 | 228
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Caucasian/White | 130 | 254 | 384
  Race: Black | 6 | 14 | 20
  Race: Asian/Oriental | 30 | 53 | 83
  Race: Other | 1 | 7 | 8
  Ethnicity: Hispanic | 40 | 94 | 134
  Ethnicity: Non Hispanic | 127 | 234 | 361
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8.37 (0.84) | 8.42 (0.88) | 8.40 (0.87)
2-Hour Postprandial Plasma Glucose (PPG) [Mean (Standard Deviation); unit: mmol/L] — The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Number of patients analyzed = 153 and 302 for Placebo and Lixisenatide treatment arms, respectively.
  mmol/L | 16.11 (3.86) | 16.47 (4.30) | 16.35 (4.15)
Average 7-Point Self Monitored Plasma Glucose (SMPG) [Mean (Standard Deviation); unit: mmol/L] — Patients recorded a 7-point plasma glucose profile before and 2 hours after each meal and at bedtime once in a week and the average value for the 7-time points was calculated. Number of patients analyzed = 155 and 301 for Placebo and Lixisenatide treatment arms, respectively.
  mmol/L | 10.58 (2.69) | 10.76 (2.61) | 10.70 (2.64)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 8.05 (2.65) | 8.13 (2.83) | 8.10 (2.76)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 88.94 (20.84) | 87.10 (20.01) | 87.72 (20.29)
Total Insulin Dose [Mean (Standard Deviation); unit: units per day] | 57.73 (34.54) | 53.43 (33.89) | 54.88 (34.14)
Glucose Excursion [Mean (Standard Deviation); unit: mmol/L] — Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the meal test, before study drug administration. Number of patients analyzed = 153 and 301 for Placebo and Lixisenatide treatment arms, respectively.
  mmol/L | 7.32 (3.43) | 7.59 (3.60) | 7.50 (3.54)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 12.43 (6.33) | 12.48 (7.04) | 12.46 (6.80)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated by dividing body weight by the height squared.
  kilogram per square meter (kg/m^2) | 32.56 (6.32) | 31.91 (6.17) | 32.13 (6.22)
Basal Insulin Treatment Duration [Mean (Standard Deviation); unit: years] | 3.20 (3.96) | 3.06 (3.37) | 3.11 (3.57)
Number of Patients With Insulin Therapy at Baseline [Number; unit: participants] — NPH included isophane insulin and insulin human injection, isophane. Premix insulin included Novolin 70/30 mix and Humalog 75/25 mix.
  participants
    Glargine | 83 | 165 | 248
    Detemir | 19 | 24 | 43
    Neutral protamine hagedorn (NPH) | 64 | 134 | 198
    Premix (Mixed Insulin) | 3 | 5 | 8
Number of Patients With Metformin use at Baseline [Number; unit: participants]
  Yes | 131 | 261 | 392
  No | 36 | 67 | 103
Metformin Daily Dose [Mean (Standard Deviation); unit: milligram (mg) per day] — Here, number of patients analyzed = 131 and 261 for Placebo and Lixisenatide treatment arm, respectively as only these participants received metformin.
  milligram (mg) per day | 2008.02 (441.88) | 1961.02 (459.07) | 1976.72 (453.38)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: Absolute change = HbA1c value at Week 24 minus HbA1c value at baseline. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population:all randomized patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures. LOCF was used. Number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo.
- Lixisenatide: 2-step initiation regimen of lixisenatide.
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 158 | 304
percentage of hemoglobin | -0.38 (0.107) | -0.74 (0.090)
Statistical Analysis 1: Comparison: Placebo vs Lixisenatide; To detect a difference of 0.5% (or 0.4%) in change from baseline to Week 24 in HbA1c between lixisenatide and placebo, 300 patients in lixisenatide arm and 150 in placebo arm would provide a power of 96% (or 86%) assuming common standard deviation of 1.3% with a 2-sided test at 5% significance level; Test type: Superiority or Other; p = 0.0002, ANCOVA — Statistical testing: 2-sided at significance level=0.05. Analysis of co-variance (ANCOVA) included treatment arms, randomization strata of screening HbA1c (<8.0, >=8.0%), metformin use (yes, no), country as fixed effects, baseline HbA1c as covariate; To control type I error, a step-down procedure described by Hochberg and Tomhane was applied; Least squares (LS) mean difference = -0.36, 95% CI 2-sided [-0.550 to -0.174], Standard Error of Mean 0.096

2. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Plasma Glucose (PPG) at Week 24
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using last observation carried forward (LOCF). Here, number of patients analyzed = patients with baseline and at least 1 post-baseline 2-hour PPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 123 | 235
mmol/L | -1.72 (0.543) | -5.54 (0.468)

3. Secondary Outcome: Change From Baseline in Average 7-Point Self Monitored Plasma Glucose (SMPG) Profiles at Week 24
Description: Patients recorded a 7-point plasma glucose profile measured before and 2 hours after each meal and at bedtime once in a week and the average value for the 7-time points was calculated. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline 7-point SMPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 153 | 294
mmol/L | -0.61 (0.238) | -1.49 (0.201)

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 1 day after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 163 | 317
mmol/L | -0.55 (0.281) | -0.63 (0.233)

5. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 161 | 311
kilogram | -0.52 (0.293) | -1.80 (0.246)

6. Secondary Outcome: Change From Baseline in Total Insulin Dose at Week 24
Description: Change was calculated for total insulin dose by subtracting the baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline total insulin dose assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: units per day
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 165 | 325
units per day | -1.93 (1.589) | -5.62 (1.317)

7. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 24
Description: The on-treatment period for this efficacy variable is time from the first dose of study drug and up to 3 days after the last dose of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 158 | 304
percentage of participants | 12.0 | 28.3

8. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than or Equal to 6.5% at Week 24
Description: as for outcome 7
Time Frame: Week 24
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 158 | 304
percentage of participants | 3.8 | 14.5

9. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy During Main 24-Week Period
Description: Routine fasting SMPG and central laboratory FPG (and HbA1c after week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after week 12) were performed. Threshold values - from baseline to Week 8: fasting SMPG/FPG >270 milligram/deciliter (mg/dL) (15.0 mmol/L), from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 24: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c > 8.5%. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 166 | 327
percentage of participants | 7.2 | 5.8

10. Other Pre Specified Outcome: Change From Baseline in Glucose Excursion at Week 24
Description: Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the standardized meal test, before study drug administration. Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is time from the first dose of study drug and up to last dosing day of study drug, on or before Visit 12 (Week 24) or Day 169 if Visit 12 is not available, and before the introduction of rescue therapy. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Missing data was imputed using LOCF. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline glucose excursion assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 123 | 233
mmol/L | -0.34 (0.469) | -4.14 (0.408)

11. Other Pre Specified Outcome: Percentage of Patients With at Least 5% Weight Loss From Baseline at Week 24
Description: as for outcome 7
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 161 | 311
percentage of participants | 3.1 | 13.2

12. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration for up to 125 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 167 | 328
participants
  Symptomatic hypoglycemia | 65 | 138
  Severe symptomatic hypoglycemia | 1 | 7

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration for up to 125 weeks
Description: Median exposure to study treatment was 560 and 559 days in lixisenatide and placebo treatment arms, respectively. The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Arm/Group | Placebo | Lixisenatide
Serious Adverse Events (participants affected / at risk) | 17/167 | 46/328
Other Adverse Events (participants affected / at risk) | 104/167 | 245/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=167) | Lixisenatide (N=328)
Anogenital warts (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Coxsackie viral infection (Infections and infestations) | 0 | 1
Incision site cellulitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Pneumonia viral (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Lens dislocation (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Retinopathy haemorrhagic (Eye disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 4 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Leriche syndrome (Vascular disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 4
Sudden cardiac death (General disorders) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Coronary angioplasty (Surgical and medical procedures) | 2 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 2 | 1
Coronary revascularisation (Surgical and medical procedures) | 1 | 0
Victim of crime (Social circumstances) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=167) | Lixisenatide (N=328)
Bronchitis (Infections and infestations) | 13 | 22
Influenza (Infections and infestations) | 9 | 28
Nasopharyngitis (Infections and infestations) | 21 | 32
Upper respiratory tract infection (Infections and infestations) | 6 | 24
Urinary tract infection (Infections and infestations) | 6 | 21
Hypoglycaemia (Metabolism and nutrition disorders) | 68 | 138
Dizziness (Nervous system disorders) | 11 | 26
Headache (Nervous system disorders) | 17 | 41
Tremor (Nervous system disorders) | 6 | 18
Hypertension (Vascular disorders) | 9 | 17
Diarrhoea (Gastrointestinal disorders) | 10 | 37
Dyspepsia (Gastrointestinal disorders) | 1 | 17
Nausea (Gastrointestinal disorders) | 16 | 96
Vomiting (Gastrointestinal disorders) | 2 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 24
Asthenia (General disorders) | 10 | 18
Blood glucose decreased (Investigations) | 7 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.